CLINICAL TRIAL: NCT03027336
Title: Randomized Controlled Clinical Trial for Assessing Tolerability and Effectiveness of Formula Coleosoma 29 in Patients With Dyslipidemia
Brief Title: Efficacy and Tolerability of the Nutraceutical Formulation Coleosoma in Dyslipidemic Subjects
Acronym: Coleosoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: DOC generici srl (Unknown)
Responsible Party: Principal Investigator, Alessandra Dei Cas, Research Assistant, MD, PhD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLEOSOMA 29-06
Record Dates: First submitted 2017-01-12; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Dyslipidemias
Keywords: dyslipidemia; dietary supplement
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: The study included two arms: a treatment arm with dietary supplement (Coleosoma) and a placebo arm.
  Coleosoma is the name of a new patented dietary supplement composed by Berberin 200 mg, Fermented Red Rice from Monascus purpureus 100 mg (correspondiing at 3 mg of monacolin K), Chitosan 100 mg e Q10 Coenzyme10 mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coleosoma (Experimental): coleosoma 500mg tablet daily
  Interventions: Dietary Supplement: Coleosoma
- placebo (Placebo Comparator): placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coleosoma — patients will take one tablet of 500mg daily for 12 weeks. No dose titration is foreseen.
  Other Names: TegraDOC
  Arms: coleosoma
Dietary Supplement: Placebo — patients will take one tablet daily for 12 weeks.
  Arms: placebo

SUMMARY:
The overall objective of the study is to assess the efficacy of Coleosoma formulation (fermented red rice, berberine and chitosan) in reducing non-HDL cholesterol in dyslipidemic patients.

DETAILED DESCRIPTION:
The incidence of cardiovascular diseases related to atherosclerosis is the leading cause of death in industrialized countries and in many developing countries. It becomes, therefore, essential to implement preventive strategies with lifestyle changes in order to prevent / control the risk factors related to cardiovascular disease.

Dyslipidemia is characterized by qualitative and quantitative alterations of plasma lipids and lipoproteins. In subjects where it is not yet indicated a statin therapy, the guidelines recommend a lifestyle (diet and exercise) act to control cardiovascular risk factors.

The formulation Coleosoma is a supplement composed of fermented red rice, berberine and chitosan. Aim of the study is to evaluate the effectiveness of coleosoma formulation in reducing non-HDL cholesterol (Non-HDL-C), which provides a measure of the cholesterol content in all atherogenic particles.

This is a single-center, randomized (3:1) and controlled double-blind phase II study that involve dyslipidemic patients with non-HDL cholesterol levels ≥ 160 mg / dl.

The study included a maximum of 4 visits for all subjects enrolled. All eligible patients at V0 (screening) undergo baseline assessments (V1) and have been allocated according to the procedure of randomization to one of the study arms. Follow-up (FU) visits for all subjects was at 4 (V2) and at 12 weeks (V3) after randomization.

Laboratory and diagnostic:

At each visits patients undergo: anthropometric and hemodynamic assessment: weight and height for Body Mass Index (BMI) calculation, waist circumference, blood pressure, heart rate; blood collection for metabolic/hormonal profile: fasting plasma glucose, HbA1c, insulin, glucagon, active glucagon-like peptide-1 (GLP-1), total gastric inhibitory polypeptide (GIP), total cholesterol, HDL-cholesterol, triglycerides, aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine, creatine phosphokinase (CPK), apolipoprotein (Apo) B, Apo A1, and inflammatory cytokines (IL-1, IL-6, IL-10, high-sensitivity C Reactive Protein (hsPCR), TNFalpha).

At V1 and V2 the Endothelial Progenitor Cells (EPC) number was evaluated with a cytofluorimetric assay.

Safety analysis has been conducted after 12 weeks treatment by determining ALT, CPK and estimated Glomerular filtration rate (eGFR) values.

This study has been sponsored by DOC generici s.r.l.

ELIGIBILITY:
Inclusion Criteria:

* non-HDL cholesterol ≥ 160 mg/dl;
* providing their written Informed Consent;
* capable of understanding the nature, purpose and study procedures

Exclusion Criteria:

* diabetes (ADA criteria)
* reduced renal (GFR<60 mL/min/1.73m2) or hepatic (transaminase levels >2.5 folds the upper reference limit) function;
* present or past history of alcohol or drug abuse
* cerebro-vascular and neoplastic diseases in the 5 years prior to study visit
* use of drugs or food supplements interfering with cholesterol levels
* pregnancy or breastfeeding;
* monogenic dyslipidemia;
* participation in other clinical trials in the previous 30 days;
* uncompensated hypothyroidism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline values of non-HDL cholesterol (mg/dl) after 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the non-HDL cholesterol value compared to baseline in the 2 arms.

SECONDARY OUTCOMES:
change from baseline values of non-HDL cholesterol (mg/dl) at 4 weeks of coleosoma treatment vs placebo | 4 weeks
  Difference in the non-HDL cholesterol value compared to baseline in the 2 arms.
change from baseline values of Free Plasma Glucose (mg/dl) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the Free Plasma Glucose value compared to baseline in the 2 arms.
change from baseline values of Body Mass Index (Kg/m2) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the BMI value compared to baseline in the 2 arms.
change from baseline values of waist circumference (cm) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the waist circumference value compared to baseline in the 2 arms.
Change from baseline values of HbA1C (%) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the HbA1C value compared to baseline in the 2 arms.
Change from baseline values of LDL Cholesterol, triglycerides and HDL cholesterol at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in theLDL Cholesterol, triglycerides and HDL cholesterol value compared to baseline in the 2 arms.
  All these parameters have the same Units of Measure (mg/dl)
Change from baseline values of ApoB/Apo A1 ratio at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the ApoB/Apo A1ratio compared to baseline in the 2 arms.
Change from baseline values of inflammatory cytokines (IL-1, IL6, IL-10, hsPCR, TNFalpha ) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the inflammatory cytokines value compared to baseline in the 2 arms.
  All these parameters have the same Units of Measure (pg/ml)
Change from baseline values of insulin (pmol/l) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the insulin value compared to baseline in the 2 arms.
Change from baseline values of hormone profile (glucagon, active GLP-1 and GIP) at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the hormone profile compared to baseline in the 2 arms. All these parameters have the same Units of Measure (pg/ml)
Change from baseline values of Endothelial Progenitor Cells (EPC) number at 12 weeks of coleosoma treatment vs placebo | 12 weeks
  Difference in the EPC number compared to baseline in the 2 arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Dei Cas, MD, Principal Investigator — University of Parma
Locations (1):
- Endocrinology Unit, Parma, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- [Background] Boekholdt SM, Arsenault BJ, Mora S, Pedersen TR, LaRosa JC, Nestel PJ, Simes RJ, Durrington P, Hitman GA, Welch KM, DeMicco DA, Zwinderman AH, Clearfield MB, Downs JR, Tonkin AM, Colhoun HM, Gotto AM Jr, Ridker PM, Kastelein JJ. Association of LDL cholesterol, non-HDL cholesterol, and apolipoprotein B levels with risk of cardiovascular events among patients treated with statins: a meta-analysis. JAMA. 2012 Mar 28;307(12):1302-9. doi: 10.1001/jama.2012.366. PMID 22453571
- [Background] El Harchaoui K, van der Steeg WA, Stroes ES, Kuivenhoven JA, Otvos JD, Wareham NJ, Hutten BA, Kastelein JJ, Khaw KT, Boekholdt SM. Value of low-density lipoprotein particle number and size as predictors of coronary artery disease in apparently healthy men and women: the EPIC-Norfolk Prospective Population Study. J Am Coll Cardiol. 2007 Feb 6;49(5):547-53. doi: 10.1016/j.jacc.2006.09.043. Epub 2007 Jan 22. PMID 17276177
- [Background] Roura S, Galvez-Monton C, Bayes-Genis A. The challenges for cardiac vascular precursor cell therapy: lessons from a very elusive precursor. J Vasc Res. 2013;50(4):304-23. doi: 10.1159/000353294. Epub 2013 Jul 9. PMID 23860201
- [Background] Vasa M, Fichtlscherer S, Aicher A, Adler K, Urbich C, Martin H, Zeiher AM, Dimmeler S. Number and migratory activity of circulating endothelial progenitor cells inversely correlate with risk factors for coronary artery disease. Circ Res. 2001 Jul 6;89(1):E1-7. doi: 10.1161/hh1301.093953. PMID 11440984
- [Background] Hill JM, Zalos G, Halcox JP, Schenke WH, Waclawiw MA, Quyyumi AA, Finkel T. Circulating endothelial progenitor cells, vascular function, and cardiovascular risk. N Engl J Med. 2003 Feb 13;348(7):593-600. doi: 10.1056/NEJMoa022287. PMID 12584367
- [Background] Dei Cas A, Spigoni V, Franzini L, Preti M, Ardigo D, Derlindati E, Metra M, Monti LD, Dell'Era P, Gnudi L, Zavaroni I. Lower endothelial progenitor cell number, family history of cardiovascular disease and reduced HDL-cholesterol levels are associated with shorter leukocyte telomere length in healthy young adults. Nutr Metab Cardiovasc Dis. 2013 Mar;23(3):272-8. doi: 10.1016/j.numecd.2011.04.005. Epub 2011 Aug 6. PMID 21824757
- [Background] Dei Cas A, Spigoni V, Ardigo D, Pedrazzi G, Franzini L, Derlindati E, Urbani S, Monti L, Gnudi L, Zavaroni I. Reduced circulating endothelial progenitor cell number in healthy young adult hyperinsulinemic men. Nutr Metab Cardiovasc Dis. 2011 Jul;21(7):512-7. doi: 10.1016/j.numecd.2009.11.011. Epub 2010 Mar 15. PMID 20227256
- [Background] Spigoni V, Lombardi C, Cito M, Picconi A, Ridolfi V, Andreoli R, Anelli N, Gnudi L, Goldoni M, Zavaroni I, Raddino R, Dei Cas A. N-3 PUFA increase bioavailability and function of endothelial progenitor cells. Food Funct. 2014 Aug;5(8):1881-90. doi: 10.1039/c3fo60641d. PMID 24942553
- [Background] Akhter J. The American Diabetes Association's Clinical Practice Recommendations and the developing world. Diabetes Care. 1997 Jun;20(6):1044-5. doi: 10.2337/diacare.20.6.1044b. No abstract available. PMID 9167126
- [Background] Pugliese G, Solini A, Bonora E, Orsi E, Zerbini G, Giorgino F, Cavalot F, Pontiroli AE, Baroni MG, Morano S, Nicolucci A, Penno G. The Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation provides a better definition of cardiovascular burden associated with CKD than the Modification of Diet in Renal Disease (MDRD) Study formula in subjects with type 2 diabetes. Atherosclerosis. 2011 Sep;218(1):194-9. doi: 10.1016/j.atherosclerosis.2011.04.035. Epub 2011 May 6. PMID 21612781
- [Background] Sola R, Valls RM, Puzo J, Calabuig JR, Brea A, Pedret A, Morina D, Villar J, Millan J, Anguera A. Effects of poly-bioactive compounds on lipid profile and body weight in a moderately hypercholesterolemic population with low cardiovascular disease risk: a multicenter randomized trial. PLoS One. 2014 Aug 1;9(8):e101978. doi: 10.1371/journal.pone.0101978. eCollection 2014. PMID 25084280